CLINICAL TRIAL: NCT07318155
Title: A Phase 2a Randomized, Double-Blind, Placebo-Controlled, Sequential Cohort Study to Evaluate the Pharmacodynamics, Safety and Pharmacokinetics of Subcutaneously Administered SRSD107 in Participants With Chronic Coronary and/or Peripheral Arterial Disease
Brief Title: A Study of SRSD107 in Participants With Chronic Coronary and/or Peripheral Arterial Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sirius Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRSD107-202
Record Dates: First submitted 2025-12-07; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease (CAD); Peripheral Arterial Disease
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SRSD107 dose level 1 (Experimental): Administered S.C.
  Interventions: Drug: SRSD107
- SRSD107 dose level 2 (Experimental): Administered S.C.
  Interventions: Drug: SRSD107
- SRSD107 dose level 3 (Experimental): Administered S.C.
  Interventions: Drug: SRSD107
- SRSD107 dose level 4 (Experimental): Administered S.C.
  Interventions: Drug: SRSD107
- Placebo (Placebo Comparator): Administered S.C.
  Interventions: Drug: 0.9 % sodium chloride

INTERVENTIONS:
Drug: SRSD107 — Administered S.C.
  Arms: SRSD107 dose level 1; SRSD107 dose level 2; SRSD107 dose level 3; SRSD107 dose level 4
Drug: 0.9 % sodium chloride — Administered S.C.
  Arms: Placebo

SUMMARY:
The study is a Phase 2a, randomized, double-blind, placebo-controlled, sequential cohort study to evaluate the pharmacodynamics (PD), safety and pharmacokinetics (PK) of multiple doses of SRSD107 in participants with coronary arterial disease (CAD) and/or peripheral arterial disease (PAD) with aspirin as background concomitant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
* Males or females aged 18 to 75 years, inclusive.
* Body mass index (BMI) between 18.0 and 35.0 kg/m2, inclusive.
* History of chronic coronary and/or peripheral arterial disease

Exclusion Criteria:

* Known bleeding disorder
* Severe heart failure with known left ventricular ejection fraction <35%, or New York Heart Association (NYHA) class III or IV symptoms.
* Genetic cardiomyopathies or other non-ischemic cardiomyopathies that are not related to atherosclerotic cardiovascular disease.
* History of ethanol abuse or addictive drug use (cannabis products allowed) within 6 months of screening.
* Receipt of an investigational drug (IP) within 30 days or 5 half-lives of that drug, whichever is longer, prior to dose administration in this study.
* Previous use of SRSD107.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in time-averaged FXI antigen | 72 weeks

SECONDARY OUTCOMES:
Percent change from baseline in FXI antigen, FXI activity and aPTT | 72 weeks
Maximal concentration of SRSD107 | 72 weeks
Area under the concentration-time curve from time 0 to infinity of SRSD107 | 72 weeks
Time to the maximal concentration of SRSD107 | 72 weeks
Incidence of adverse events | 72 weeks

IPD SHARING:
Plan to Share IPD: No